CLINICAL TRIAL: NCT06772116
Title: Jupiter Registry: Prospective Registry for Patients Undergoing Focal Therapy for Localized Prostate Cancer
Brief Title: Focal Therapy in Localized Prostate Cancer: a Prospective Registry
Acronym: JR
Status: Not yet recruiting | Type: Observational
Sponsor: Institut Mutualiste Montsouris (Other)
Collaborators: European Association of Urology Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: JUPITER2024
Record Dates: First submitted 2024-12-27; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Prostate; Prostate Cancer
Keywords: Focal Therapy; HIFU; Cryotherapy; FLA; Focal Brachytherapy; IRE; VTP; RFA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with intermediate-risk prostate cancer: he study includes patients with intermediate-risk prostate cancer (PCa), as defined by the European Association of Urology (EAU) risk groups, and a life expectancy of more than 10 years. Eligible patients must have undergone both targeted and systematic biopsies confirmed through the US-MRI fusion technique. All participants are required to provide informed, written consent before being included in the study.
  Interventions: Procedure: Focal Therapy

INTERVENTIONS:
Procedure: Focal Therapy — Primary focal treatment (targeted or partial gland ablation) of PCa lesion(s) detected on mpMRI, where a PCa ISUP 2 or 3 has been identified (PCa ISUP 1 outside the treatment areas is acceptable, regardless of volume).
  Focal treatment will be performed using one of the following energy-based techniques: high-intensity focused ultrasound (HIFU), cryotherapy (CRYO), brachytherapy (BT), irreversible electroporation (IRE), focal laser ablation (FLA), vascular-targeted photodynamic therapy (VTP), or radiofrequency ablation (RFA). The specific technique will depend on the rules, approvals, and regulations of the country where the treatment is performed.
  Other Names: Targeted Therapy for Prostate Cancer; Partial Gland Ablation (PGA); Energy-Based Ablative Therapy

SUMMARY:
The principal aim of the registry is to collect data on focal therapy (FT) for the treatment of intermediate-risk prostate cancer across Europe. Data will be gathered on cancer absence following treatment, survival rates, and the absence of disease failure or progression. Information will be collected from as many centers as possible over the next 5 years to enhance understanding of when focal therapy should be used, which energy types are most effective, and how patients respond to treatment, including its side effects and impact on quality of life.

This Europe-wide data collection will contribute to improving care by informing the development of enhanced national and international guidelines for prostate cancer treatment with focal therapy.

DETAILED DESCRIPTION:
Focal Therapy has been introduced and evaluated as a minimally invasive treatment aimed at improving management strategies for localized prostate cancer. This technique consists of ablating the dominant lesion while preserving as much of the non-cancerous tissue as possible, and treating only the areas that require intervention.

The aim of the Jupiter Registry is to establish a registry for patients with intermediate-risk prostate cancer undergoing FT. The registry will prospectively gather standardized data from multiple European centers.

The goal is to collect data from as many centers as possible over a 5-year follow-up period to inform clinical practices on FT indications, energy type selection, and patient outcomes, including efficacy, complications, and quality of life. This Europe-wide, reliable data will help develop national and international recommendations and guidelines to improve patient care.

This registry will subsequently enable the development of Jupiter Studies, a series of registry-based studies designed to analyze specific research questions regarding focal therapy in patients with intermediate-risk prostate cancer. The aim is to generate robust evidence on various aspects (efficacy, safety, functional impact, oncological impact) of focal therapy in a real-world evidence context.

Data such as PSA levels, MRI results, and biopsy outcomes will be collected during patient follow-up.

Additionally, data on salvage treatments will be documented, including the type and complications of any salvage treatments performed during follow-up up to 60 months post-FT.

Although the registry provides a uniform data collection on the population of patients with intermediate-risk localized prostate cancer who have undergone FT in accordance with EMA recommendations (Guideline on registry-based studies EMA/426390/2021), the principal and secondary aims defined below will subsequently enable the realization of the Jupiter Studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with intermediate risk PCa based on EAU risk groups with life expectancy > 10 years
* Prior targeted + systematic biopsy using US-MRI fusion technique
* Primary focal treatment (targeted or partial gland ablation) of PCa lesion(s) detected on mpMRI, where PCa ISUP 2 or 3 has been identified. PCa ISUP 1 outside the treatment areas is acceptable, regardless of volume.
* Focal treatment was performed using one of the following energies: high-intensity focused ultrasound (HIFU), cryotherapy (CRYO), brachytherapy (BT), irreversible electroporation (IRE), focal laser ablation (FLA), vascular-targeted Photodynamic (VTP) and radiofrequency ablation (RFA) according to the country rules, approvals, and regulations of each country in which they are applied. The registry cannot be used as a clinical trial or post-marketing surveillance study of the technologies applied.
* Free, informed and written consent

Exclusion Criteria:

* Patients with intermediate risk treated with focal therapy without a previous targeted + systematic prostate biopsy with US-MRI fusion technique.
* Primary focal treatment of PCa ISUP 2 or 3 in areas of prostate without evidence of lesions on MRI (MRI-invisible prostate cancer)
* Patients with histological diagnosis of PCa with ISUP > 1 outside the areas of treatment
* Primary whole gland treatments using ablative energy HIFU, cryotherapy, IRE, FLA, VTP and/or RFA
* Primary subtotal/total treatments using ablative energy HIFU, cryotherapy, IRE, FLA, VTP and/or RFA
* Life expectancy <10 years
* Previous treatment of PCa (excluded a period of Active Surveillance)
* High risk PCa based on EAU risk groups.
* Locally advanced PCa
* Metastatic hormone-sensitive prostate cancer (mHSPC)
* Metastatic castration-resistant prostate cancer (mCRPC)
* Non-Metastatic Castration-Resistant Prostate Cancer (nmCRPC)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study includes patients with intermediate-risk prostate cancer (PCa), as defined by the European Association of Urology (EAU) risk groups, with a life expectancy of more than 10 years. The criteria for intermediate-risk PCa are: PSA 10-20 ng/mL or GS 7 (ISUP grade 2/3) or cT2b (based on digital rectal examination).
  According to the latest EAU guidelines, patients with low-risk localized prostate cancer (PCa) should be offered active surveillance, while those with high-risk localized PCa should receive multimodal treatment. For intermediate-risk patients, alongside prostatectomy and radiotherapy, the EAU guidelines strongly recommend "focal ablative therapy within clinical trials or registries."
  The indication for treatment with focal therapy is entrusted to the clinicians of each center.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2032-02 (Estimated)

PRIMARY OUTCOMES:
Rate of Negative Histological Findings for Prostate Cancer (PCa) on Target-Guided Biopsy of the Treated Area | 12 months
  The rate of negative histological findings for PCa (any ISUP grade) on target-guided biopsy of the treated area at 12 months post-FT (target or partial gland ablation) among patients who underwent biopsy (for any reason) among the cohort of 1,000 patients with intermediate-risk PCa enrolled.

SECONDARY OUTCOMES:
Overall Survival (OS) | 12-, 24-, 36-, 48- and 60-months after FT treatment
  Time from the date of focal therapy (FT) to the date of death from any cause.
Cancer-Specific Survival (CSS) | 12-, 24-, 36-, 48-, and 60-months after FT treatment
  The time from the date of focal therapy (FT) to the date of death due to prostate cancer.
Metastasis-Free Survival (MFS) | 12-, 24-, 36-, 48-, and 60-months after FT treatment
  The time from the date of focal therapy (FT) to the date of the first imaging-confirmed distant metastasis.
FT Impact on Erectile Function | Baseline and at 12 months after FT treatment (optional: every 12 months until 60 months post-treatment)
  Changes from baseline to 12 months after FT in erectile function, as measured by the Sexual Health Inventory for Men (SHIM). SHIM is a validated 5-item questionnaire with a total score ranging from 1 to 25, where higher scores indicate better erectile function.
  The questionnaire is included in the "Functional Assessment" (FA) and will be administered throughout the entire follow-up period.
FT Impact on Lower Urinary Tract Symptoms | Baseline and at 12 months after FT treatment (optional: every 12 months until 60 months post-treatment)
  Changes from baseline to 12 months after FT in urinary symptoms, as measured by the International Prostate Symptoms Score (IPSS). IPSS is a validated 7-item questionnaire with a total score ranging from 0 to 35, where higher scores indicate more severe urinary symptoms.
  The questionnaire is included in the "Functional Assessment" (FA) and will be administered throughout the entire follow-up period.
FT impact on Ejaculatory Function | Baseline and at 12 months after FT treatment (optional: every 12 months until 60 months post-treatment)
  Changes from baseline to 12 months after FT in ejaculatory function, as measured by the 1st and 4th items of the Male Sexual Health Questionnaire-Ejaculatory Dysfunction Short Form (MSHQ-EjD SF). Scores for the 1st item range from 0 to 5, with higher scores indicating better ejaculatory function. Scores for the 4th item range from 0 to 5, with higher scores indicating greater bother related to ejaculatory dysfunction as perceived by the patient.
  The questionnaire is in included in the "Functional Assessment" (FA) and will be used during the whole follow-up.
FT impact on Quality of Life | Baseline and at 12 months after FT treatment (optional: every 12 months until 60 months post-treatment)
  Changes from baseline to 12 months after FT in quality of life related to prostate cancer, as measured by the Overall Prostate Cancer QoL Score of the Expanded Prostate Cancer Index Composite for Clinical Practice (EPIC-CP). Scores range from 0 to 100, with higher scores indicating worse quality of life.
  The questionnaire is in included in the "Functional Assessment" (FA) and will be used during the whole follow-up.
Complications | at 3, 6, 9, and 12 months, and then annually until 60 months after treatment.
  Complications related to the FT treatments will be recorded using a text-free module that includes the option to select specific types of common complications (e.g., untreated bacteriuria, urinary tract infection (UTI) treated with antibiotics, acute urinary retention, bleeding, pain not relieved by common painkillers, or severe hematoma). In all cases, the Clavien-Dindo classification will be applied to categorize any post-operative complications recorded.
Prostate Failure-Free Survival (pFFS) | 12-, 24-, 36-, 48- and 60-months after FT treatment
  Time from the date of focal therapy until the occurrence of an ISUP 2 PCa or higher in the treated area and/or untreated area found during the follow up.
  The success of FT is evaluated based on the absence of clinically significant prostate cancer throughout the entire prostate (prostate-based approach). The presence of clinically significant prostate cancer in either the untreated and/or treated areas will be considered a failure.
Area Treated Failure-Free Survival (aFFS) | 12-, 24-, 36-, 48- and 60-months after FT treatment
  "Time from the date of focal therapy until the occurrence of an ISUP 2 PCa or higher in the treated area, as identified during follow-up. The success of FT is evaluated based solely on the treated area (area-treated-based approach), and only the presence of clinically significant prostate cancer within the treated area will be considered a failure.
Progression free survival (PFS) | 12-, 24-, 36-, 48- and 60-months after FT treatment
  Will be calculated using the time from the date of focal therapy (FT) to the date progression is reported. Progression is defined as the requirement for whole-gland treatments, including salvage radical prostatectomy, salvage external beam radiotherapy, salvage brachytherapy, salvage whole gland ablation, and systemic therapy (androgen deprivation therapy, chemotherapy, anti-androgens, PARP inhibitors, AKT inhibitors, immune checkpoint inhibitors, and radiopharmaceutical therapy).
Salvage Treatments Rate | 12-, 24-, 36-, 48- and 60-months after FT treatment
  The rate of salvage treatments, including Active Surveillance, Watchful Waiting strategy, Salvage Radical Prostatectomy, Salvage External Beam Radiotherapy, Salvage Brachytherapy, Salvage Whole Gland Ablation, and Systemic Therapies (e.g., androgen deprivation therapy, chemotherapy, anti-androgens, PARP inhibitors, AKT inhibitors, immune checkpoint inhibitors, and radiopharmaceutical therapy), will be recorded for each patient.
Rate of complications associated with Salvage Treatments | at 3, 6, 9, and 12 months, and then annually until 60 months after treatment.
  Complications associated with Salvage Treatments will be recorded using a text-free module that includes the option to select specific types of common complications (e.g., untreated bacteriuria, urinary tract infection (UTI) treated with antibiotics, acute urinary retention, bleeding, pain not relieved by common painkillers, or severe hematoma). In all cases, the Clavien-Dindo classification will be applied to categorize any post-operative complications recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Barret, MD, PhD, Principal Investigator — Institut Mutualiste Montsouris; Juan I Martinéz-Salamanca, MD, PhD, Principal Investigator — Lyx Institute of Urology

IPD SHARING:
Plan to Share IPD: No
Local Research Institutions may also use the data that entered in the database for further research, if their research project has been validated by the Scientific Committee. Local Research Institutions may export their data themselves using the exporting tool in Excel, CSV or SPSS format for data. In this case, Research Institutions access the data in the database and undertake to only use these data for the purposes of the research project that has been validated.
  During the entire duration of the Jupiter Registry the data will remain pseudonymized in Castor EDC (cool-down period). During this timeframe data is kept in a protected state or with restricted access before it is made available for further analysis or actions such as anonymization or permanent deletion.
  At the end of Jupiter registry, EAU-RF will anonymize the Study Data according to Regulations and to actual official European guidelines and create a "Data haven" ensuring that it is impossible to re-identify the data.

REFERENCES:
- [Background] Lebastchi AH, George AK, Polascik TJ, Coleman J, de la Rosette J, Turkbey B, Wood BJ, Gorin MA, Sidana A, Ghai S, Tay KJ, Ward JF, Sanchez-Salas R, Muller BG, Malavaud B, Mozer P, Crouzet S, Choyke PL, Ukimura O, Rastinehad AR, Pinto PA. Standardized Nomenclature and Surveillance Methodologies After Focal Therapy and Partial Gland Ablation for Localized Prostate Cancer: An International Multidisciplinary Consensus. Eur Urol. 2020 Sep;78(3):371-378. doi: 10.1016/j.eururo.2020.05.018. Epub 2020 Jun 10. PMID 32532513
- [Background] Borkowetz A, Blana A, Bohmer D, Cash H, Ehrmann U, Franiel T, Henkel TO, Hocht S, Kristiansen G, Machtens S, Niehoff P, Penzkofer T, Pinkawa M, Radtke JP, Roth W, Witzsch U, Ganzer R, Schlemmer HP, Grimm MO, Hakenberg OW, Schostak M. German S3 Evidence-Based Guidelines on Focal Therapy in Localized Prostate Cancer: The First Evidence-Based Guidelines on Focal Therapy. Urol Int. 2022;106(5):431-439. doi: 10.1159/000521882. Epub 2022 Feb 10. PMID 35144260
- [Background] Hopstaken JS, Bomers JGR, Sedelaar MJP, Valerio M, Futterer JJ, Rovers MM. An Updated Systematic Review on Focal Therapy in Localized Prostate Cancer: What Has Changed over the Past 5 Years? Eur Urol. 2022 Jan;81(1):5-33. doi: 10.1016/j.eururo.2021.08.005. Epub 2021 Sep 4. PMID 34489140
- [Background] van der Poel HG, van den Bergh RCN, Briers E, Cornford P, Govorov A, Henry AM, Lam TB, Mason MD, Rouviere O, De Santis M, Willemse PM, van Poppel H, Mottet N. Focal Therapy in Primary Localised Prostate Cancer: The European Association of Urology Position in 2018. Eur Urol. 2018 Jul;74(1):84-91. doi: 10.1016/j.eururo.2018.01.001. Epub 2018 Jan 17. PMID 29373215